CLINICAL TRIAL: NCT06347484
Title: Developing a Learning COmmunity to Increase eNgagemeNt and Enrollment in Cardiovascular Clinical Trials
Brief Title: Developing a Learning COmmunity to Increase eNgagemeNt and Enrollment in Cardiovascular Clinical Trials (CONNECT)
Acronym: CONNECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Morgan State University (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00411716
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Hypertension; Diabetes Type 2; Stroke; Recruitment; Overweight and Obesity; Hyperlipidemias
Keywords: Recruitment; Diversity; Inclusion; Clinical Trials; Cardiovascular Disease; Community Engagement; Registry; Digital Health
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus, Type 2; Stroke; Overweight; Obesity; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Participants enrolling in CONNECT will receive tailored educational text messages and opportunities to join cardiovascular research studies. Recruitment will occur via electronic health record (EHR)-informed and community-engaged methods. Enrollment yield will be evaluated for all outreach modalities, both overall and by priority populations (women and Black and Latino adults). The study will also assess participant trust in biomedical research, awareness of clinical trials, and willingness to participate at baseline, 6 months, and 12 months.
  Sub-study 1: This sub-study will evaluate the effectiveness of three EHR-informed outreach methods: patient portal message, email, and postal mail. Potentially eligible individuals will be identified through EHR query and randomly assigned to one of these methods. Enrollment yield will be assessed by outreach method and priority population.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Educational Text-Messages and Connection to Cardiovascular Research Opportunities (Experimental): All participants who enroll in CONNECT, regardless of method of contact, will receive educational text messages and connection to cardiovascular research opportunities.
  Interventions: Behavioral: Educational Text-Messages and Connection to Cardiovascular Research Opportunities
- EHR-Informed Recruitment Sub-Study #1, Arm #1: Contact Method, Patient Portal Message (Active Comparator): Potential participants will be identified using an EHR query and will be randomized to receive a recruitment message via the patient portal message. This message will invite the participant to join CONNECT.
  Interventions: Behavioral: EHR-informed Recruitment Method of Contact
- EHR-Informed Recruitment Sub-Study #1, Arm #2: Contact Method, Email (Active Comparator): Potential participants will be identified using an EHR query and will be randomized to receive a recruitment message via email. This message will invite the participant to join CONNECT.
  Interventions: Behavioral: EHR-informed Recruitment Method of Contact
- EHR-Informed Recruitment Sub-Study #1, Arm #3: Contact Method, Postal Mail (Active Comparator): Potential participants will be identified using an EHR query and will be randomized to receive a recruitment message via postal mail. This message will invite the participant to join CONNECT.
  Interventions: Behavioral: EHR-informed Recruitment Method of Contact

INTERVENTIONS:
Behavioral: EHR-informed Recruitment Method of Contact — The intervention being studied here is the method of contact (patient portal vs. email vs. postal mail) after being identified in the EHR
  Arms: EHR-Informed Recruitment Sub-Study #1, Arm #1: Contact Method, Patient Portal Message; EHR-Informed Recruitment Sub-Study #1, Arm #2: Contact Method, Email; EHR-Informed Recruitment Sub-Study #1, Arm #3: Contact Method, Postal Mail
Behavioral: Educational Text-Messages and Connection to Cardiovascular Research Opportunities — All participants who enroll in CONNECT, regardless of method of contact, will receive educational text messages and connection to cardiovascular research opportunities. Text messages will be tailored and include content on cardiovascular health promotion and research participation.
  Arms: Educational Text-Messages and Connection to Cardiovascular Research Opportunities

SUMMARY:
The CONNECT: "Developing a learning COmmunity to increase eNgagemeNt and Enrollment in cardiovascular Clinical Trials" is comprehensive, participant-centered learning platform designed to increase diversity in cardiovascular disease research among women and Black and Latino adults. CONNECT will deploy electronic health record (EHR)-informed and community-engaged recruitment approaches to identify and recruit adults with cardiovascular disease or a cardiovascular disease risk factor to join CONNECT. Participants who join CONNECT will receive tailored educational information on cardiovascular health and research participation via text message. Participants will also have the opportunity to be connected to ongoing cardiovascular research studies based on basic demographic information and areas of interest. The educational information will be sent to participants for 12 months. The CONNECT platform will be used to evaluate recruitment methods. The investigators hypothesize the proportion of women and Black and Latin adults enrolled in trials that partner with CONNECT will be higher following the use of CONNECT for recruitment. Investigators also hypothesize that participating in CONNECT will increase participants' clinical trial awareness, trust, and willingness to participate in clinical trials.

DETAILED DESCRIPTION:
The CONNECT project, titled "Developing a learning COmmunity to increase eNgagemeNt and Enrollment in cardiovascular Clinical Trials," seeks to establish an comprehensive learning platform aimed at improving diversity and representation in cardiovascular research. It encompasses three primary objectives:

1. Identifying best practices for research recruitment and engagement among women and Black and Latino adults.
2. Increasing participation in cardiovascular health research among women and Black and Latino adults.
3. Improving trust in and awareness of cardiovascular research among women and Black and Latino adults.

A multi-method recruitment campaign will be implemented, utilizing both electronic health record (EHR)-informed and community-based strategies. A sub-study will be conducted to understand the effectiveness of EHR-informed recruitment. This sub-study will randomly assign a subsample of individuals identified in the EHR to one of three outreach modalities: patient portal message, email, and postal mail. Enrollment yield will be calculated for each recruitment method, with logistic regression modeling estimating the odds of enrollment by recruitment outreach type, both overall and among different demographic groups.

Upon enrollment, participants will specify preferences for receiving text messages regarding heart health, research education, and study opportunities. Messaging will focus on cardiovascular health prevention, management strategies, and research processes, with the aim of fostering trust in research within the community. Pre-post surveys will be distributed to assess changes in clinical trial awareness, trust in medical research, and willingness to participate in trials at baseline, 6 months, and 12 months post-enrollment. Interaction terms will be used to evaluate differences in outcomes by race, ethnicity, and sex.

The process for matching participants to research within the CONNECT project involves individual researchers submitting requests to the CONNECT study team for access to the learning community as a recruitment resource, followed by approval Institutional Review Board (IRB) approval. Upon access, researchers can retrieve, and view records of participants matched to respective studies, ensuring access only to data pertinent to the research objectives. Verification of IRB approval is mandated, and the CONNECT study team will request documentation from the individual research team's IRB to confirm compliance before granting access. Researchers using CONNECT must document eligibility and enrollment data for each CONNECT participant matched to the participants study. Proportions of participants matched to and enrolled in ongoing research studies will be tabulated and compared across demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years or older
* Residing in the US
* Self-identifies as having cardiovascular disease or cardiovascular risk factors
* Has a mobile phone and is willing to receive text-messages
* Can read in English or Spanish

Exclusion Criteria:

* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Participant accrual by priority population | Baseline
  The total number of participants enrolled in CONNECT, divided by the total number recruited. This will be completed for each recruitment method (EHR-Informed vs. Community-Engaged)
Participant accrual by recruitment method | Baseline
  The total number of participants enrolled in CONNECT, divided by the total number recruited. This will be completed for each priority population (women, Black, and Latino Adults).

SECONDARY OUTCOMES:
Participant accrual in partnering cardiovascular research studies | Baseline, 6-months, and 12-months
  The proportion of CONNECT participants who enroll into a cardiovascular research study.
Trust in Biomedical Research using the Perceptions of Research Trustworthiness Scale (PoRT) | Baseline, 6-months, and 12-months
  Trust in biomedical research among participants will be assessed using an 18-item instrument, the Perceptions of Research Trustworthiness Scale (PoRT). Possible scores range from 1 (Definitely Disagree) to 5 (Definitely Agree), with 1 indicating higher trust and 5 indicating lower trust.
Clinical trials awareness and knowledge will be assessed using items adapted from the Health Information National Trends Survey (HINTS) | Baseline, 6-months, and 12-months
  Awareness of clinical trials will be assessed by asking participants, "Have you ever heard of a clinical trial?" with response options including "Yes," "No," or "Don't Know." While level of knowledge about clinical trials will be assessed by asking participants to describe level of knowledge about clinical trials, with response options including "I don't know anything about clinical trials," "I know a little bit about clinical trials," and "I know a lot about clinical trials."
Willingness to participate in research will be measured by asking participants one related question | Baseline, 6-months, and 12-months
  Participants will be asked, "In the future, if you developed a health problem like heart disease, would you consider joining a clinical trial that was testing a new heart disease treatment that could help you?" Response options include: "I would not participate," "I might participate," "I probably would participate," "I definitely would participate," and "Not sure/haven't thought about it."

CONTACTS AND LOCATIONS:
Overall Officials: Hailey N Miller, PhD, RN, Principal Investigator — Johns Hopkins School of Nursing; Cheryl R Dennison Himmelfarb, PhD, RN, ANP, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Miller HN, Wong E, Byiringiro S, Hussain Z, Guerrero Vazquez M, Lewis-Land C, Skelton B, Curriero S, Foster A, Moghimi F, Tomiwa O, Shaia J, Sheikhattari P, Wang NY, Dennison Himmelfarb CR. CONNECT Platform to Increase Diverse Engagement and Enrollment in Cardiovascular Clinical Research: Rationale, Design, and Lessons Learned in Early Implementation. J Am Heart Assoc. 2025 Aug 19;14(16):e038351. doi: 10.1161/JAHA.124.038351. Epub 2025 Aug 12. PMID 40792590